CLINICAL TRIAL: NCT07007039
Title: Remote Therapeutic Monitoring: Pilot Implementation-Effectiveness Study
Brief Title: Pilot Remote Therapeutic Monitoring in Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Miriam Rafferty, Director of Implementation Science, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00217608
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: exercise; activity tracking; rehabilitation; remote monitoring
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Therapeutic Monitoring (Other): Participants will receive 3 months of remote therapeutic monitoring via a connected health app and personal activity tracker to monitor their physical activity and exercise behaviors.
  Interventions: Other: Datos Health App

INTERVENTIONS:
Other: Datos Health App — Tracking participants step activity, workout frequency, minutes in target heart rate zone, and/or strength bouts completed over 3 month period. Individualized goals will be selected and set with a customized amount by a rehabilitation provider with at least monthly follow up contact to modify goals.

SUMMARY:
The goal of this clinical trial is to learn about exercise and physical activity in individuals who are undergoing cancer treatment. The clinical trial is embedded in a pilot implementation feasibility study. The main implementation questions it aims to answer are to understand the implementation feasibility, acceptability and appropriateness of remote monitoring from providers and participants. The main clinical trial outcomes are to explore the effectiveness of remote therapeutic monitoring to achieve individual goal attainment related to exercise defined as number of daily steps, weekly exercise minutes, strength sessions or decreased physical activity variability.

During the course of the study: Participants will use activity trackers and a mobile phone application to monitor their exercise participation over 3 months.

DETAILED DESCRIPTION:
The study aims to evaluate the implementation and clinical effectiveness of Remote Therapeutic Monitoring (RTM) in cancer rehabilitation. RTM is a reimbursable tool that enables clinicians (physical therapists, occupational therapists, and physicians) to remotely monitor adherence to exercise and physical activity (PA), addressing barriers such as limited time and energy for in-person appointments during cancer treatment. We will implement three months of RTM in 20 individuals undergoing or within six months of chemotherapy, immunotherapy, or cell therapy. We will evaluate the following aims:

1. Implementation Outcomes: Assess RTM's feasibility, acceptability, appropriateness, sustainability, and satisfaction from the perspectives of therapists, physicians, and patients using validated questionnaires and interviews.

2: Clinical Trial Outcomes: Measure RTM's effectiveness in achieving patient-centered goals, such as increasing or maintaining exercise, PA, strength training, or energy conservation, and its impact on quality of life using PROMIS-29+2.

The findings will inform future large-scale research and enhance cancer rehabilitation outcomes by improving accessibility and personalized care through RTM integration.

ELIGIBILITY:
Inclusion Criteria:

* Are ambulatory as their primary means of mobility without an assistive device except for single point cane or walking sticks in community
* Have a diagnosis of cancer (undergoing chemo, radiation, surgery, immunotherapy, or cell therapy (transplants and Chimeric Antigen Receptor t-cell therapy (CAR-T)) or in cancer survivorship
* Participating in Outpatient rehabilitation services at time of enrollment, or recommended by physician for participation in study
* Have a goal to increase or maintain physical activity (e.g., steps per day or minutes of moderate to vigorous exercise per week) or strength bouts - personal goal and willingness to address physical activity
* Have a smart phone
* Willing to accept Datos' Terms and Conditions

Exclusion Criteria:

* o Individuals with cognitive or communication disorders (including dementia) which would limit their ability to interact with the RTM in this pilot phase

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Metric 1 | Daily, through study completion, average 3 months
  steps per day
PROMIS 29+2 | completed at baseline and at study completion, average of 3 months
  A self report survey used to assess health report quality of life. It contains 31 total questions.

SECONDARY OUTCOMES:
Physical Activity Metric 2 | Daily, through study completion, average 3 months
  minutes of exercise in target heart rate zone
Physical Activity Metric 3 | weekly, through study completion, average 3 months
  Number of strength training bouts

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Rafferty, PT, DPT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheville AL, Moynihan T, Herrin J, Loprinzi C, Kroenke K. Effect of Collaborative Telerehabilitation on Functional Impairment and Pain Among Patients With Advanced-Stage Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):644-652. doi: 10.1001/jamaoncol.2019.0011. PMID 30946436
- [Background] da Silva HEC, Santos GNM, Ferreira Leite A, Mesquita CRM, de Souza Figueiredo PT, Miron Stefani C, de Santos Melo N. The feasibility of telehealth in the monitoring of head and neck cancer patients: a systematic review on remote technology, user adherence, user satisfaction, and quality of life. Support Care Cancer. 2022 Oct;30(10):8391-8404. doi: 10.1007/s00520-022-07109-z. Epub 2022 May 6. PMID 35524146
- [Background] Schmitz KH, Campbell AM, Stuiver MM, Pinto BM, Schwartz AL, Morris GS, Ligibel JA, Cheville A, Galvao DA, Alfano CM, Patel AV, Hue T, Gerber LH, Sallis R, Gusani NJ, Stout NL, Chan L, Flowers F, Doyle C, Helmrich S, Bain W, Sokolof J, Winters-Stone KM, Campbell KL, Matthews CE. Exercise is medicine in oncology: Engaging clinicians to help patients move through cancer. CA Cancer J Clin. 2019 Nov;69(6):468-484. doi: 10.3322/caac.21579. Epub 2019 Oct 16. PMID 31617590
- [Background] Stout NL, Santa Mina D, Lyons KD, Robb K, Silver JK. A systematic review of rehabilitation and exercise recommendations in oncology guidelines. CA Cancer J Clin. 2021 Mar;71(2):149-175. doi: 10.3322/caac.21639. Epub 2020 Oct 27. PMID 33107982
- [Background] Ficarra S, Thomas E, Bianco A, Gentile A, Thaller P, Grassadonio F, Papakonstantinou S, Schulz T, Olson N, Martin A, Wagner C, Nordstrom A, Hofmann H. Impact of exercise interventions on physical fitness in breast cancer patients and survivors: a systematic review. Breast Cancer. 2022 May;29(3):402-418. doi: 10.1007/s12282-022-01347-z. Epub 2022 Mar 12. PMID 35278203
- [Background] Malone S, Prewitt K, Hackett R, Lin JC, McKay V, Walsh-Bailey C, Luke DA. The Clinical Sustainability Assessment Tool: measuring organizational capacity to promote sustainability in healthcare. Implement Sci Commun. 2021 Jul 17;2(1):77. doi: 10.1186/s43058-021-00181-2. PMID 34274004
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Rosebrock K, Sinn M, Uzunoglu FG, Bokemeyer C, Jensen W, Salchow J. Effects of Exercise Training on Patient-Specific Outcomes in Pancreatic Cancer Patients: A Scoping Review. Cancers (Basel). 2023 Dec 18;15(24):5899. doi: 10.3390/cancers15245899. PMID 38136443